CLINICAL TRIAL: NCT02065804
Title: Trigger-point Blockade in Persistent Pain After Laparoscopically Assisted Groin Hernia Repair
Brief Title: Trigger-point Blockade in Persistent Pain After Laparoscopical Groin Hernia Repair
Acronym: Trigger-lap
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, mads u werner, MD, DMSc, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-3-2011-130-lap
Record Dates: First submitted 2014-02-15; First posted 2014-02-19 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Chronic Pain
Keywords: Herniorrhaphy; Surgical Equipment; Chronic Pain; Inguinal Herniorrhaphy; Laparoscopy; Surgical Outcome
MeSH Terms: conditions — Chronic Pain | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active drug (Experimental): 10 ml of bupivacaine 2.5 mg/ml deposited by ultra-sound guidance around the spermatic cord
  Interventions: Drug: Bupivacaine
- Placebo (Placebo Comparator): 10 ml of normal saline deposited by ultra-sound guidance around the spermatic cord
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — injection, once, 5 min
  Other Names: Bupivacain "SAD"; 0.9% Sodium-chloride

SUMMARY:
Groin hernia repair is a common procedure performed in approximately 2,000 patients per one million inhabitants. Severe chronic pain following groin hernia repair is seen in 2-5% of the patients indicating that a large number of patients each year suffer from debilitating reduction in health-related quality of life.

This study examines the effect of ultra-sound guided blocks with local anesthesia in the groin in regard to pain relief and sleep quality.

The hypothesis of the study is that a block will confer significant pain relief to patients with severe chronic pain following laparoscopical groin hernia repair.

DETAILED DESCRIPTION:
This placebo-controlled, randomized, double-blind, cross-over study in subjects with severe pain after laparoscopically assisted groin hernia repair, examines the effect of an ultra-sound guided local anesthetic block of a trigger-point, situated near the spermatic cord at the superficial inguinal ring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent pain (< 6 mo) after laparoscopical groin hernia repair
* Patients with maximal pain area 3 cm or less from the superficial inguinal ring
* Patients living in the Capital Region of Denmark (Region Hovedstaden) or the Region of Zealand (Region Sjælland)

Exclusion Criteria:

* Known allergy to bupivacaine or other local anesthetics of amide-type
* Declared incapable of making his/hers own affairs
* Does not comprehend Danish in writing or speech
* Cognitive impairment to a degree influencing the testing reliability
* Known recurrence of the inguinal hernia
* Other surgical procedures performed in the groin or on the external genitals
* Neuropathy affecting the groin region caused by other conditions, e.g. post-stroke, multiple sclerosis, herniated intervertebral disc
* Abuse of alcohol or drugs
* Unable to cooperate with the sensory examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Normalized summed pain intensity differences (SPID) | 20 min
  The number of patients with normalized summed pain intensity differences (SPID) of more or equal to 50% after bupivacaine AND SPID less or equal to 25% after placebo.

SECONDARY OUTCOMES:
Thermal thresholds | 20 min
  Quantitative changes in thermal thresholds (warmth detection threshold, cool detection thresholds, heat pain threshold) after bupivacaine compared to placebo
Suprathreshold heat stimulation | 20 min
  Quantitative changes in pain rating to suprathreshold heat stimulation after bupivacaine compared to placebo
Pressure pain thresholds | 20 min
  Quantitative changes in pain rating to pressure algometry stimulation after bupivacaine compared to placebo
Sensory mapping | 20 min
  Quantitative changes in area of cool hypoesthesia assessed by a thermal roller after bupivacaine compared to placebo
Pain questionnaire | 7 days
  Quantitative changes in summed pain intensity differences (SPIDs) assessed morning and evening after bupivacaine compared to placebo
Sleep quality questionnaire | 7 days
  Quantitative changes in sleep quality assessed each morning after bupivacaine compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Mads Werner, Principal Investigator — Multidisciplinary Pain Center, Neuroscience Center, Rigshospitalet, Copenhagen University Hospital, DENMARK; Henrik Kehlet, MD, DMSc, Study Chair — Section of Surgical Pathophysiology, Juliane Marie Center, Copenhagen University Hospital, DENMARK
Locations (1):
- Multidisciplinary Pain Center, Neuroscience Center, Copenhagen University Hospital, DENMARK, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be submitted as supplementary material in the final manuscript

REFERENCES:
- [Background] Linderoth G, Kehlet H, Aasvang EK, Werner MU. Neurophysiological characterization of persistent pain after laparoscopic inguinal hernia repair. Hernia. 2011 Oct;15(5):521-9. doi: 10.1007/s10029-011-0815-z. Epub 2011 Apr 9. PMID 21479588